CLINICAL TRIAL: NCT00562575
Title: A Randomised, Double-blind, Placebo Controlled Study to Evaluate the Pharmacodynamics, Safety, Tolerability and Pharmacokinetics Profile of SLx-4090 Over 14 Days Dosing in Subjects With High Triglyceride Values
Brief Title: Evaluation of Safety and Effects of SLx-4090 After Dosing for 14 Days in Subjects With High Triglycerides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLx-4090-07-03
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — 6-(4'-trifluoromethyl-6-methoxybiphenyl-2-ylcarboxamido)-1,2,3,4-tetrahydroisoquinoline-2-carboxylic acid phenyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SLx-4090
  Interventions: Drug: SLx-4090
- 2 (Placebo Comparator): Matching Placebo Dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLx-4090
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose is to investigate the effect of oral doses of SLx-4090 over 14 days on subjects with high triglycerides.

DETAILED DESCRIPTION:
1. Serum triglycerides
2. Serum lipids and lipoproteins
3. Safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with high triglyceride levels
* Male or female subjects between age 18 and 65 years, inclusive

Exclusion Criteria:

* History of drug abuse
* Any prescribed or over the counter medication taken within 2 weeks prior to administration of study drug or within 6 times the elimination half-life
* Blood donation of more than 500ml blood in the previous 3 months
* Any confirmed significant allergic reaction against any drug or multiple allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Serum triglycerides | 14 days

SECONDARY OUTCOMES:
Adverse events and vital signs | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Grit Anderson, MD, Principal Investigator — FOCUS clinical Drug Development GmbH
Locations (1):
- FOCUS Clinical Drug Development GmbH, Neuss, Germany